CLINICAL TRIAL: NCT01331161
Title: Systems Biology of Zoster Vaccine (ZOSTAVAX®) in Young and Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Nadine Rouphael, MD, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00050285; U19AI090023 (NIH); HIPCVAX005 (Other: Other)
Record Dates: First submitted 2011-04-06; First posted 2011-04-07 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-01

CONDITIONS: Shingles
Keywords: shingles vaccine; immune responses
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Older group (Experimental): Participants between the ages of 60-79
  Interventions: Biological: ZOSTAVAX
- Younger group (Experimental): Participants between the ages of 25-40
  Interventions: Biological: ZOSTAVAX

INTERVENTIONS:
Biological: ZOSTAVAX — shingles vaccine, one dose
  Other Names: shingles vaccine

SUMMARY:
Vaccination is the most effective way of preventing infectious diseases. Despite the success of vaccines in general, vaccines induce diminished antibody responses and lower protection in the elderly in particular. This could be explained by a defect in the early responses of an ageing immune system. A better understanding of the basic immunological mechanisms that mediate vaccine efficacy is incomplete. Such information is critical and could greatly decrease both the cost and the time to new vaccine development particularly for the geriatric population.

In this trial, the investigators will study the immunologic differences of the FDA approved licensed shingles vaccine between a younger and an older group. Thirty three healthy volunteers between the ages of 25-40 and forty four healthy volunteers between the ages of 60-79 will be enrolled in the study. Each participant in the study will be given one shingles shot. Blood work will be obtained one month before vaccination, on the day of vaccination, one day, three days, seven days, fourteen days, one month, three months and six months after vaccination. Throughout the duration of the study, the participants will be monitored for safety.

DETAILED DESCRIPTION:
RATIONALE: Zoster vaccine is known to induce diminished antigen-specific T cell responses and lower protection in the elderly. Here we hypothesize that this is due to intrinsic defects in innate responses to the live attenuated virus, which translates into sub-optimal functional adaptive immune responses. Therefore, early innate signatures of vaccination should correlate with, and predict the immunogenicity of Zoster vaccine in the young and elderly.

STUDY DESIGN: Double center, open label study in which adult healthy volunteers will be vaccinated with Zoster vaccine. Blood samples will be collected on day D-30 (pre- vaccination) D0 (at vaccination) and D1, D3, D7, D14, D30, D90 and D180 (post vaccination) to study innate and adaptive immunity responses. Even though Zoster vaccine is considered safe, volunteers are asked to report and record any local or systemic AEs for 7 days post-vaccination. Also AEs will be reported for 30 days post-vaccination any SAE for 180 days post vaccination. AEs developing the day of the blood draw will also be reported

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and give informed consent.
* Immunocompetent subjects aged 25-40 years, or community dwelling subjects between the ages of 60-79.

Exclusion Criteria:

* Young adults aged 25-40 years who are Varicella-Zoster virus seronegative or equivocal results (mean value OD for Varicella-Zoster virus IgG lower than 1.1 by commercial enzyme-linked immunosorbent assay (ELISA) (Hope Clinic: IgG VZV ELISAII-Wampole Laboratories®, NJ, USA- Vaccine Research Trials Center:: Liaison VZV IgG Assay, DiaSorin, Italy)
* Receipt of immune products:

  * Receipt of blood products within 6 months prior to vaccination with Zoster vaccine or expected receipt through 6 months after vaccination with Zoster vaccine*
  * Receipt of any vaccine within 4 weeks prior to vaccination with Zoster vaccine or expected receipt within 4 weeks after vaccination with Zoster vaccine*
  * Receipt of Zoster vaccine or varicella vaccines at any time prior to study entry.
* Subject taking any non-topical antiviral therapy with activity against herpes viruses, including but not limited to acyclovir, famciclovir, valacyclovir, and ganciclovir 3 days prior to vaccination or 14 days after*.
* Prior history of shingles.
* Presence of certain co morbidities or immunosuppressive states such as:

  * Chronic medical problems including (but not limited to) insulin-dependent diabetes, severe heart, lung, liver, or kidney diseases; auto immune diseases; severe gastrointestinal diseases; and uncontrolled hypertension.
  * Alcohol or drug abuse and psychiatric conditions that in the opinion of the investigator would preclude compliance with the trial or interpretation of safety or endpoint data.
  * Impaired immune function or chronic infections including (but not limited to) HIV, hepatitis B or C, tuberculosis, organ transplant, cancer, current and or expected receipt of chemotherapy, radiation therapy, steroids [i.e., > 20 mg of prednisone given daily or on alternative days for 2 weeks or more in the past 90 days*); (nasal and topical steroids are allowed)],antitumor necrosis factor agents, or any other immunosuppressive therapy, anatomic or functional asplenia, congenital immunodeficiency.
  * Pregnant or breast-feeding women, or women expecting to conceive 30 days before and 90 days after vaccination**.
* Conditions that could affect the safety of the volunteers such as:

  * Severe reactions to prior vaccinations.
  * History of anaphylactic/anaphylactoid reaction to gelatin, neomycin or any other component of the vaccine. Neomycin allergy manifested as contact dermatitis is not a contraindication to receiving this vaccine.
  * History of bleeding disorders
* Any acute illness, including any fever (> 100.4 F [> 38.0C], regardless of the route) within 3 days prior to study entry *.
* Social, occupational, or any other condition that in the opinion of the investigator might interfere with compliance with the study and vaccine evaluation.

Note:

*An individual who initially is excluded from study participation based on one or more of the time-limited exclusion criteria (e.g., acute illness, receipt or expected receipt of live or inactivated vaccines ) may be considered for enrollment once the condition has resolved as long as the subject continues to meet all other entry criteria.

Subjects receiving > 20 mg/day of prednisone or its equivalent daily or on alternate days for more than 2 weeks may enter the study after therapy has been discontinued for more than 3 months.

**Women of child-bearing potential (not surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy or who are not postmenopausal for ≥1 year) must agree to practice adequate contraception that may include, but is not limited to, relationship with vasectomized partner, barrier methods such as condoms, diaphragms, spermicides, intrauterine devices, and licensed hormonal methods for 30 days before and 90 days after zoster vaccination.

Ages: 25 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-07; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Rouphael, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - University of Colorado, Aurora, Colorado
  - Emory University, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from Atlanta and Denver from July 2011 until March 2012 using flyers
Period: Overall Study
Arm/Group | Older Group | Younger Group
Started | 44 | 33
Completed | 43 | 31
Not Completed | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Age 60-79 Years: Participants between the ages of 60-79 years received a single dose of the Zoster vaccine (ZOSTAVAX®) subcutaneously.
- Age 25-40 Years: Participants between the ages of 25-40 years received a single dose of the Zoster vaccine (ZOSTAVAX®) subcutaneously.
- Total: Total of all reporting groups
Arm/Group | Age 60-79 Years | Age 25-40 Years | Total
Number analyzed (Participants) | 44 | 33 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 33 | 53
  >=65 years | 24 | 0 | 24
Age, Continuous [Median (Full Range); unit: years] | 68 [60 to 77] | 33 [25 to 40] | 61 [25 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 48
  Male | 19 | 10 | 29
Region of Enrollment [Number; unit: participants]
  United States | 44 | 33 | 77
Ethnicity [Number; unit: Participants]
  Hispanic | 3 | 3 | 6
  Non hispanic | 41 | 30 | 71

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Innate Immunity Signatures That Correlate With the T Cell Adaptive Immunity Responses After ZOSTAVAX
Description: The primary outcomes will identify the number of participants with innate immunity signatures in the young and older groups that correlate with the T cell adaptive immunity responses after ZOSTAVAX
Time Frame: 2 years
Population: participants with immunoglobulin gene responses that correlated with adaptive immune responses
Measure: Number; unit: participants
Groups:
- Participants 60-79 Years: participants who received one dose of vaccine
- Participants 25-40 Years of Age: participants with one dose of vaccine
Arm/Group | Participants 60-79 Years | Participants 25-40 Years of Age
Number analyzed (Participants) | 44 | 33
participants | 44 | 33

2. Secondary Outcome: The Number of Participants With Innate Immune Signatures That Correlate With the B and T Cells Adaptive Immunity Responses After ZOSTAVAX
Description: The number of participants with innate immune signatures in the young and old groups that correlate with the B and T cells adaptive immunity responses after ZOSTAVAX
Time Frame: 2 years
Population: Participants with both T and B cell responses to vaccine
Measure: Number; unit: participants
Arm/Group | Age 60-79 Years | Age 25-40 Years
Number analyzed (Participants) | 44 | 33
participants | 23 | 27

ADVERSE EVENTS:
Arm/Group | Older Group | Younger Group
Serious Adverse Events (participants affected / at risk) | 2/44 | 0/33
Other Adverse Events (participants affected / at risk) | 13/44 | 3/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Older Group (N=44) | Younger Group (N=33)
Hyponatremia (Endocrine disorders) | 1 (1) | 0 (0) — resulted in hospitalization- unrelated to study product
Breast Cancer (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Breast cancer unrelated to study product
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Older Group (N=44) | Younger Group (N=33)
Local Injection site reactions (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0) — All were attributed as related to study product- severity was between 1 and 2- all resolved
Bruise at blood draw site (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) — realted to phlebotomy intervention- all resolved
Cold symptoms (Infections and infestations) | 3 (3) | 2 (2) — None related to study product- severity varied between 1 to 3 - all resolved

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No